CLINICAL TRIAL: NCT04591977
Title: HPV Self-sampling Among Women at Penn State Hershey Well Women Appointments
Brief Title: Self-Sampling for Human Papillomavirus (HPV) at Well Women Appointments
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment, preliminary analysis indicates that primary endpoint has been met
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer L. Moss, PhD, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14033
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: HPV
Keywords: HPV; Cervical Cancer; Self-Sampling; Cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants who enroll in the study will be asked to complete an HPV self-sampling test in addition to attending their well-woman visit and receiving a clinician-sampled Pap Smear/HPV test. Participants will collect the sample at home and mail it back to the Penn State Health clinical laboratory, where the results will be compared to those obtained from the Pap Smear/HPV test at their clinic appointment. Participants will also complete a follow up survey over the phone after their sample is collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Self-Sampling Kit (Experimental): Self-Sampling kit (Evalyn Brush) to collect samples for analysis for HPV/Cervical cancer screening.
  Interventions: Device: HPV Self-Sampling Kit (Evalyn Brush)

INTERVENTIONS:
Device: HPV Self-Sampling Kit (Evalyn Brush) — The Evalyn Brush is a self-sampling kit that can be used to collect a sample to screen for HPV/Cervical cancer at home.

SUMMARY:
This study seeks to compare the accuracy and acceptability of Human Papillomavirus (HPV) testing self-sampling kit versus standard clinician-sampled HPV testing for cervical cancer screening. The primary outcome of this study is the concordance between screening results on self-sampling kits compared to clinician-collected HPV test and Pap smear results. Secondary endpoints will include acceptability of self-sampling and barriers to cervical cancer screening. These endpoints will be analyzed to try to circumvent barriers to the cervical cancer screening and ascertain whether self-sampling is a viable alternative to clinician sampling.

DETAILED DESCRIPTION:
The American Cancer Society estimates that 4,170 women in the United States (US) will die from cervical cancer in 2018. Screening can reduce cancer mortality by (1) detecting malignancies when they are more treatable and (2) for some tests, identifying precancerous lesions for removal. Guidelines recommend cytology and/or human papillomavirus (HPV) testing for cervical cancer screening among women ages 30-65 years, but screening rates are suboptimal.

To help bridge these gaps in screening, HPV self-sampling would be an alternative to clinical screening. However, there are concerns about the comparability and acceptability of self-sampling kits. The impact of the proposed project is to compare HPV self-screening results with Pap smear results and clinician-collected HPV tests to ultimately improve the uptake of HPV screening. This study will be conducted in a normal risk population.

Subjects who have an upcoming well-woman appointment will be identified from Penn State Health, Department of Family and Community Medicine, clinic schedules. Clinicians who are a part of the study team will identify these patients two weeks prior to their appointment and send their information to a study coordinator, who will then call these patients to provide more information and assess their interest in participating. Patients who schedule within the two week period or were not contacted by a study team member for any reason will be given a card with general information about the study at their well-woman visit so that these women can contact a study team member if they are interested. A total of 197 participants will be recruited into this study.

Interested participants will be screened for eligibility over the phone and sent a self-sampling kit through the mail with a Summary Explanation of Research form, instructions, and pre-paid mailer to return the kit. Participants may collect their sample two weeks before or after their well-woman visit. A study team member will contact the participants at different time points within the 28 day window to determine whether the sample was collected and to administer the follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 Years
* Penn State Health, Family and Community Medicine, patient attending a well-woman visit
* Able to collect the sample within two weeks of visit
* Female
* Intact cervix
* Speaks, reads, or writes in English

Exclusion Criteria:

* Pregnancy
* Cognitively Impaired
* Incarcerated
* Complete hysterectomy
* History of cervical treatment for abnormal Pap/HPV test (cryotherapy, LEEP)

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Moss, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Shieh Y, Eklund M, Sawaya GF, Black WC, Kramer BS, Esserman LJ. Population-based screening for cancer: hope and hype. Nat Rev Clin Oncol. 2016 Sep;13(9):550-65. doi: 10.1038/nrclinonc.2016.50. Epub 2016 Apr 13. PMID 27071351
- [Background] U. S. Preventive Services Task Force. Final recommendation statement: Cervical cancer: Screening; 2018. https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/cervical-cancer-screening2. Accessed 2018.
- [Background] Saslow D, Solomon D, Lawson HW, Killackey M, Kulasingam SL, Cain J, Garcia FA, Moriarty AT, Waxman AG, Wilbur DC, Wentzensen N, Downs LS Jr, Spitzer M, Moscicki AB, Franco EL, Stoler MH, Schiffman M, Castle PE, Myers ER; ACS-ASCCP-ASCP Cervical Cancer Guideline Committee. American Cancer Society, American Society for Colposcopy and Cervical Pathology, and American Society for Clinical Pathology screening guidelines for the prevention and early detection of cervical cancer. CA Cancer J Clin. 2012 May-Jun;62(3):147-72. doi: 10.3322/caac.21139. Epub 2012 Mar 14. PMID 22422631
- [Derived] Wong A, Morgis R, Entenman J, Ramirez SI, Hays AL, Wright TS, Scartozzi CM, Ruffin MT, Moss JL. Exploratory Analysis of Concordance Between Clinician-Collected and Self-Sampled Human Papillomavirus Tests in a Small Cohort of Average- and High-Risk Patients. Womens Health Rep (New Rochelle). 2024 Mar 13;5(1):259-266. doi: 10.1089/whr.2024.0004. eCollection 2024. PMID 38516651

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants in this group were those scheduled for routine cervical cancer screening.
Period: Overall Study
Arm/Group | Participants
Started | 46
Completed | 35
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
annual household income [Count of Participants; unit: Participants]
  < $50,000 | 4
  $50,000+ | 29
  unknown/not reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Concordance of Screening Results of the Self-sampling Kit Compared to Clinical-collected Samples
Description: Number of participants whose results of the self-sampling kit were in concordance with the clinician-sampled HPV test and clinician-sampled Pap smear results.
Time Frame: Within two weeks of the well-woman visit
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 35
Participants | 35

2. Secondary Outcome: Number of Completed Self-Sampling Kits
Description: The number of participants provided a kit vs. those who completed the sample collection
Time Frame: 28 days (two weeks before or after the well-woman visit)
Population: Total number of participants that were provided with a self-sampling kit.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Sampling Kit
Number analyzed (Participants) | 46
Participants | 35

3. Secondary Outcome: Number of Participants Who Reported Problems With Using Self-Sampling Kits
Description: The number of participants, among those who completed the sample collection, who reported problems using the self-sampling kit.
Time Frame: Within two weeks of the well-woman visit
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 35
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over 41 days, which was the longest period between the clinician-collected and self-collected tests.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

LIMITATIONS AND CAVEATS:
small sample size due to slow participant accrual, exclusion of patients who do not seek care (population most likely to benefit from self-sampling)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT04591977/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT04591977/ICF_003.pdf